CLINICAL TRIAL: NCT00401596
Title: A Multicenter, Randomized, Controlled, Open-Label Study to Evaluate the Safety of Xolair in Moderate to Severe Persistent Asthma Subjects Already Treated With Other Therapies (ALTO)
Brief Title: A Study to Evaluate the Safety of Xolair in Moderate to Severe Persistent Asthma Patients (ALTO)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: Q2143g
Record Dates: First submitted 2006-11-17; First posted 2006-11-20 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-03

CONDITIONS: Asthma
Keywords: ALTO
MeSH Terms: conditions — Asthma | interventions — Omalizumab

INTERVENTIONS:
Drug: Xolair (omalizumab)

SUMMARY:
This was a multicenter, open label, randomized, controlled, safety trial in subjects aged 6-75 years with a diagnosis of moderate to severe, persistent asthma. A total of 1899 subjects were randomized (2:1) to either the active treatment group or the control group. Upon successful completion of the screening period (~2 weeks), each subject entered the 24 week study.

ELIGIBILITY:
Inclusion Criteria:

* Documented physician diagnosis of moderate to severe, persistent asthma, defined in the National Heart, Lung, and Blood Institute (NHLBI) guidelines as FEV1 < 80% predicted for height, age, and sex or a history of FEV1 < 80%
* Between 6 and 75 years old at the time of screening (Visit 1 [Week -2])
* Current treatment with the following medications: Moderate doses of any inhaled steroid preparation on a daily basis for at least 30 days prior to screening; and/or oral steroids at a stable dose on a daily basis for at least 30 days prior to screening; and currently treated with at least one of the following drugs on a daily basis at a stable dose for at least 30 days prior to screening: long-acting β-adrenergic (salmeterol), leukotriene receptor antagonist (LTRA), xanthine derivatives, or sodium cromoglycate
* Signed informed consent (in the case of a minor, consent must have been given by the child's parent or legal guardian)
* Serum IgE level of ≥ 30 IU/mL and ≤ 1300 IU/mL and a body weight ≥ 20 kg and ≤ 150 kg and fell within the protocol-defined dosing table ranges
* For females of childbearing potential, in the opinion of the investigator, use of an effective method of contraception to prevent pregnancy and agreement to continue to practice an acceptable method of contraception for the duration of their participation in the study
* Willingness to participate fully for the duration of the study

Exclusion Criteria:

* Current active AEE defined as requiring initiation or increase in oral steroid dose or treatment with at least a doubling of inhaled steroid dose
* Thrombocytopenia as evidenced by platelets < 100,000/uL
* Pregnancy or lactation
* Previous randomization in this study
* Use of any experimental drug within 30 days prior to study screening
* Known hypersensitivity to any ingredients of Xolair, including excipients (sucrose, histidine, polysorbate 20)
* Diagnosis of aspirin or nonsteroidal anti-inflammatory drug-induced asthma
* Active lung disease other than asthma (e.g., chronic bronchitis, emphysema, cystic fibrosis, chronic obstructive pulmonary disease)
* History of smoking within 2 years of the study screening visit or history of smoking ≥ 10 pack years
* Significant systemic disease (e.g., infection, hematologic, renal, hepatic, coronary heart disease or other cardiovascular diseases, endocrinologic or gastrointestinal disease) within the previous 3 months
* History of neoplasia
* History of noncompliance to medical regimens
* Any systemic condition requiring regular administration of immunoglobulin

Ages: 6 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1899
Dates: Start 2000-07; Study Completion 2002-07 (Actual)

PRIMARY OUTCOMES:
Incidence of all serious adverse events.

SECONDARY OUTCOMES:
Incidence of all adverse events during the treatment phase of the study
Incidence of protocol defined asthma exacerbation episodes (AEEs) during the treatment phase of the study
Nocturnal symptoms as measured by the modified Inner City Asthma Study Morbidity Assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Yamo Deniz, M.D., Study Director — Genentech, Inc.

REFERENCES:
- [Derived] Busse WW, Humbert M, Haselkorn T, Ortiz B, Trzaskoma BL, Stephenson P, Garcia Conde L, Kianifard F, Holgate ST. Effect of omalizumab on lung function and eosinophil levels in adolescents with moderate-to-severe allergic asthma. Ann Allergy Asthma Immunol. 2020 Feb;124(2):190-196. doi: 10.1016/j.anai.2019.11.016. Epub 2019 Nov 22. PMID 31760132